CLINICAL TRIAL: NCT04313270
Title: Subclinical Atherosclerosis in Patients With Familial Hypercholesterolemia Treated With Evolocumab®
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Matteo Di Minno, Associate Professor of Internal Medicine, Federico II University
Other Study IDs: 2015/261
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Hypercholesterolemia, Familial
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — evolocumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with FH starting a treatment with Evolocumab®
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — 12 weeks of treatment with Evolocumab

SUMMARY:
Protein convertase subtilisin kexin type 9 (PCSK-9) inhibitors demonstrated efficacy in cholesterol reduction and in the prevention of cardiovascular events. The investigators will evaluate changes in lipid profile, oxidation markers and subclinical atherosclerosis in patients with familial hypercholesterolemia (FH) during 12 weeks of treatment with a PCSK-9 inhibitor, Evolocumab®.

DETAILED DESCRIPTION:
Several studies emphasize the role of high levels of low-density lipoprotein cholesterol (LDL-C) as the main causative factor in atherosclerosis development. Among patients with hypercholesterolemia, those with very high levels of LDL-C exhibit increased prevalence of subclinical atherosclerosis and a higher atherosclerosis progression, thus leading to a significantly higher CV risk. Endothelial dysfunction is the earliest stage of the atherosclerotic process and even a trigger of CV events. Flow-mediated dilation (FMD) is widely accepted as an accurate and non-invasive method to assess vascular reactivity and, in turn, as a surrogate marker of subclinical atherosclerosis and an independent predictor of CV events. It's well known that hypercholesterolemia has been associated with decreased endothelial function and increased oxidative stress. Although statin treatment represented for years the gold standard as lipid lowering therapy, the target LDL-C is not always achieved, mainly among patients with very high levels of LDL-C. More recently, PCSK-9 inhibitors demonstrated efficacy in LDL-C reduction, in the prevention from CV events and in atherosclerotic burden regression. Some data showed an effect of PCSK-9 inhibitors on endothelial function, but no evidence is available on effect on LDL subfractions. Small dense LDL (sd-LDL) are considered an emerging risk factor for cardiovascular disease due to a greater atherogenic potential [ ] and are important markers for predicting CV risk.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of FH (clinical and/or genetic)
* eligibility of patients to start a treatment with PCSK-9 according to 2016 ESC guidelines.

Exclusion Criteria:

* age < 18 years
* inability to understand or sign the informed consent
* high level of transaminases ( >3x upper normal limit)
* hypertriglyceridemia ( >150 mg/dl)
* end-stage renal disease (filtration rate < 30 ml/min/mq)
* current malignant disease or a diagnosis of malignancy in the 2 years prior to the first visit
* previous exposure to PCSK-9 inhibitors
* presence of hypercholesterolemia secondary to other causes (hypothyroidism, hormone therapies, corticosteroids etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients attending the lipid clinic of the Department of Clinical Medicine and Surgery, Federico II University Hospital with very high levels of LDL-C (above the 95th percentile when compared with a sex- and age-matched general population), normal triglyceride levels and presumed autosomal dominant transmission of hypercholesterolemia in the family were screened for inclusion in the present study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Subclinical atherosclerosis | 12 weeks
  evaluation of subclinical atherosclerosis in patients receiving Evolocumab

CONTACTS AND LOCATIONS:
Locations (1):
- Matteo Di Minno, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannuzzo G, Buonaiuto A, Calcaterra I, Gentile M, Forte F, Tripaldella M, Di Taranto MD, Giacobbe C, Fortunato G, Rubba PO, Di Minno MND. Association between causative mutations and response to PCSK9 inhibitor therapy in subjects with familial hypercholesterolemia: A single center real-world study. Nutr Metab Cardiovasc Dis. 2022 Mar;32(3):684-691. doi: 10.1016/j.numecd.2021.10.025. Epub 2021 Nov 11. PMID 34991937